CLINICAL TRIAL: NCT02287129
Title: Metabolic and Molecular Response Evaluation for the Individualization of Therapy in Adenocarcinomas of the Gastroesophageal Junction
Brief Title: Evaluation for the Individualization of Therapy in Adenocarcinomas of the Gastroesophageal Junction
Acronym: MEMORI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEM-0000-SIV-0028-I
Record Dates: First submitted 2014-10-07; First posted 2014-11-10 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Adenocarcinoma of the Esophagogastric Junction
Keywords: Potentially R0 - resectable AEG and primary tumor category; Histologically confirmed AEG I-III; Functional operability; Intense FDG tracer uptake of the tumor
MeSH Terms: interventions — Oxaliplatin; Epirubicin; Capecitabine; Fluorouracil; Carboplatin; Paclitaxel; Radiation; Biopsy; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Responder (Experimental): Oxaliplatin Epirubicin Capecitabine 5-FU Carboplatin Paclitaxel Radiation Biopsy
  Interventions: Drug: Oxaliplatin; Drug: Epirubicin; Drug: Capecitabine; Drug: 5-FU; Drug: Carboplatin; Drug: Paclitaxel; Radiation: radiation; Procedure: Biopsy
- Responder (Active Comparator): Oxaliplatin Epirubicin Capecitabine 5-FU Biopsy
  Interventions: Drug: Oxaliplatin; Drug: Epirubicin; Drug: Capecitabine; Drug: 5-FU; Procedure: Biopsy

INTERVENTIONS:
Drug: Oxaliplatin — 130 mg/m2
  Other Names: Oxaliplan
Drug: Epirubicin — 50 mg/m2
  Other Names: Epi Teva
Drug: Capecitabine — 625 mg/m2
  Other Names: Xeloda
Drug: 5-FU — 200 mg/m2
  Other Names: 5-FU medac
Drug: Carboplatin — 2 mg/ml min
  Other Names: Carboplatin SUN
  Arms: Non-Responder
Drug: Paclitaxel — 50 mg/m2
  Other Names: Taxomedac
  Arms: Non-Responder
Radiation: radiation — total dosage 41,4 Gy
  Other Names: intensitive neoadjuvant radiochemotherapy (INRCT)
  Arms: Non-Responder
Procedure: Biopsy — translational analysis
  Other Names: esophagogastroduodenoscopy

SUMMARY:
Metabolic and Molecular Response evaluation for the individualization of therapy in adenocarcinomas of the gastroesophageal junction by evaluation of the R0 resection rate for patients with metabolically (ie, according to PET criteria) chemotherapy-resistant locally advanced AEG, who receive an intensified neoadjuvant chemoradiotherapy (INRCT). Additonal efforts will be done by investigation of molecular and metabolic biomarkers in relation to their predictive and prognostic value by correlating them with histopathologic responses and clinical outcome in an exploratory approach.

DETAILED DESCRIPTION:
Adenocarcinomas of the esophagus and the esophagogastric junction (AEG) are clinically-topographically divided into subtypes I-III according to the Siewert classification and show an increased incidence. Neoadjuvant and/or perioperative chemotherapy or preoperative radiochemotherapy is well established in the management of AEG. However, a significant number of patients do not respond to preoperative chemotherapy, suffering from toxicity and facing a worse outcome due to lower R0 resection rates. Previous results from the MUNICON-1 and MUNICON-2 trials have shown that PET-based therapy individualization can be successfully integrated in neoadjuvant treatment algorithms.

Tumor-free resection edges (R0) constitute the greatest prognostic advantage in terms of overall survival. However, the R0 resection rates for patients who, according to early metabolic response evaluation, have not responded to the chemotherapy, have not been satisfactory, even after conversion to an - albeit moderate - radiochemotherapy in the MUNICON-2 trial. Thus, this patient population (so-called non responders) so far lack a beneficial neoadjuvant therapy modality.

Based on these results, the primary goal of MEMORI study is to evaluate the R0 resection rate for patients with metabolically (ie, according to PET criteria) chemotherapy-resistant locally advanced AEG, who receive an intensified neoadjuvant chemoradiotherapy (INRCT). Secondary it is planned to investigate molecular and metabolic biomarkers in relation to their predictive and prognostic value by correlating them with histopathologic responses and clinical outcome in an exploratory approach.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed AEG I-III
* Potentially R0 - resectable AEG and primary tumor category UT2 -4
* Functional operability : Exclusion of OP - limiting comorbidities
* Intense FDG tracer uptake of the tumor during Baseline PET/CT examination and thus suitability for monitoring and early response prediction by FDG - PET ( [ 18F ] - FDG uptake in the tumor at baseline > 1.35 x liver SUV + 2 x standard deviation of the liver SUV)
* Performance status (ECOG ) 0 or 1
* Age : ≥ 18
* creatinine clearance > 60ml/min measured in a 24 h urine or calculated with the Cockgroft -Gault formula
* bilirubin ≤ 1.5 times upper limit of normal , serum transaminases (GOT

  / GPT ) ≤ 3 times ULN
* leukocytes ≥ 3.5 g / l, platelet ≥ 100 g / l
* Negative pregnancy test (determination of beta- HCG in urine or serum) in women of childbearing potential
* A signed consent form after implementation of medical education

Exclusion Criteria:

* Existing distant metastases (M1b)
* Tumor infiltration into the tracheobronchial system
* Previous radiotherapy targeted at the thorax
* Lack of ability of the patient to adhere to the protocol rules
* Manifest heart failure despite optimal medication> NYHA I
* existing angina pectoris at rest or undergoing stress without clarification via interventional cardiology and / or myocardial infarction within the last 6 months
* Existing pregnancy or lactation
* childbearing or fertility without using recognized safe methods of contraception
* Coexisting other malignant diseases with the exception of a non-melanomatuous, localized skin tumor or carcinoma in situ of the cervix
* absence of a signed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 1 day of surgery (in between day 28 to day 43 after radio-chemotherapy)
  R0 resection rate of patients suffering from metabolically (following PET criteria) chemotherapy-resistant, locally advanced AEG, who receive a more intensive neoadjuvant radio-chemotherapy (INRCT)

SECONDARY OUTCOMES:
Regression | 1 day of surgery (in between day 28 to day 43 after radio-chemotherapy)
  Histological regression defined by Becker Criteria
Overall survival | from day 0 to follow up visit 6 (24 months after surgery)
  Overall survival defined as period from start of study to death (if necessary censored by end of follow-up period)
Disease-free survival | from day 0 to follow up visit 6 (24 months after surgery)
  Disease-free survival, defined as period from start of study to earlier occurring event: death or relapse until end of follow-up; Relapse will be separated into events of "local failure", "distant failure" and "local and distant failure"
QLQ-C30 | from day 0 to follow up visit 6 (24 months after surgery)
  Quality of life, analyzed via EORTC QLQ-C30 questionnaires
Metabilic response rate | from day 0 to one time point of time period day 14 to 28 after chemotherapy
  Metabolic response rate under neoadjuvant chemotherapy
Translational analysis | 1 day of surgery (in between day 28 to day 43 after radio-chemotherapy)
  Translational analysis for identification of tumor determinants relevant for prognosis and therapy
Adverse Events | from day 0 to follow up visit 6 (24 months after surgery)
  Occurence of AEs
QLQ-OG25 | from day 0 to follow up visit 6 (24 months after surgery)
  Quality of life, analyzed via EORTC QLQ-OG25 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jens Siveke, Prof. Dr., Principal Investigator — II. Medizinische Klinik, Klinikum rechts der Isar (MRI) der TUM,Ismaninger Str. 22
Locations (1):
- 2nd department of the Medical Clinic of the Technical University Munich, Munich, Bavaria, Germany